CLINICAL TRIAL: NCT03515174
Title: A Randomized Controlled Trial Comparing Active Intervention at Diagnosis With Usual Care to Improve the Psycho-social Care in the Adolescent and Young Adult Oncology (AYAO) Population
Brief Title: Trial Comparing Active Intervention At Diagnosis With Usual Care to Improve Psycho-social Care in AYAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/2949
Record Dates: First submitted 2018-03-28; First posted 2018-05-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma; Lymphoma; Sarcoma; Cancer
Keywords: Adolescent and Young Adult Oncology; Carcinoma; Lymphoma; Sarcoma; Cancer
MeSH Terms: conditions — Carcinoma; Lymphoma; Sarcoma; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Program (Experimental): Patients will participate in a structured supportive care program.
  Interventions: Other: Supportive Care Program; Other: Usual Care
- Control Group (Active Comparator): Patients in the control group will receive usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Supportive Care Program — This program takes place within one month post-diagnosis of cancer. It will include three info-educational session. After that, recommendations for further consultation with specific healthcare professionals will be made based on the concerns and needs of patients at baseline. Patient will also be given usual care.
  Arms: Interventional Program
Other: Usual Care — Patients will be provided with an information booklet by the study team on self-management of cancer- and treatment-related symptoms, which is routinely provided by the National Cancer Centre of Singapore (NCCS) after cancer diagnosis. Usual general advice is provided by the medical oncologists during the routine consultations.

SUMMARY:
Adolescents and young adults (AYA) patients experience significant distress in specific areas at diagnosis. The investigators hypothesize that providing developmentally-appropriate AYA-specific psychosocial care, with an individualized multi-disciplinary program will alleviate this distress, as well as improve health-related quality of life (HRQOL).

The investigators' primary aim is to evaluate the impact of psychosocial interventions on HRQOL. The secondary aims are to firstly identify the types of psychosocial distress experienced and secondly, to assess the feasibility of implementing a psychosocial screening and intervention program amongst AYA patients newly diagnosed with cancer.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 39 years old
* Newly diagnosed with any form of cancers
* Capable of giving informed consent (by patients or parents, whichever applicable)
* Ability to understand and willingness to sign a written informed consent document
* Able to speak and understand English
* Able to commit to attending the 3 info-educational sessions as well as patient-directed additional visits

Exclusion Criteria:

* Patients with uncontrolled brain metastasis.
* Patients who are unable to commit to attend all 3 info-educational sessions
* Patients who are unable to communicate in English.

Ages: 16 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Extent of symptom burden measured using Rotterdam Symptom Checklist (RSCL) | 6 months post recruitment
  The Rotterdam Symptom Checklist (RSCL) is a self-report measure to assess the quality of life of cancer patients. It uses a 4-point Likert-type scales (not at all, a little, quite a bit, very much) to measure four domains, namely the physical symptom distress (23 items), psychological distress (7 items) activity level (8 items) overall valuation of life (1 item). The higher the score, the higher the level of burden or impairment. Standardized scores of scales can also be obtained when comparing different scales by transforming raw scores into scores on a 100-point scale using the formula [(raw scale score - minimum raw score) / (maximum - minimum score)] x 100 = transformed score.
Health-related quality of life using PedsQL 4.0 Generic Core Scales | 6 months post recruitment
  Pediatrics Quality of Life Inventory (PedsQL) is a model used to measure health-related quality of life (HRQOL) in adolescents and young adults by generating a physical health summary score and psychosocial health summary score both ranging from 0-100, whereby a higher score suggests a better HRQOL. It encompasses physical, mental, and social health, the core dimensions of health defined by the World Health Organization, as well as is school functioning to generate pediatric HRQOL.

SECONDARY OUTCOMES:
Patients' distress levels using the National Comprehensive Cancer Network (NCCN) Distress Thermometer | 6 months post recruitment
  NCCN Distress Thermometer is a screening tool that measures distress on a 0 to 10 scale, whereby 0 indicates "No distress" and 10 indicates "Extreme distress". The Distress Thermometer also includes a problem checklist to identify problems that contribute to the score. These include practical problems, family problems, emotional problems, spiritual/religious concerns and physical problems that cancer patients may have.
Satisfaction Questionnaire | At 3 months from baseline
  The satisfaction questionnaire is adapted from a client satisfaction questionnaire incorporating questions about communication with healthcare providers. Patients rate their satisfaction of the info-education sessions - the way it is conducted and content and if their needs have been met on a Likert Scale. This ranges from 1 to 5: with 1 being strongly disagree and, 2 being disagree, 3 being neutral, 4 being agree and 5 being strongly agree. The total score of each individual item is summed up, with higher scores indicating a favourable response to the info-educational sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen YL Poon, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zebrack B, Isaacson S. Psychosocial care of adolescent and young adult patients with cancer and survivors. J Clin Oncol. 2012 Apr 10;30(11):1221-6. doi: 10.1200/JCO.2011.39.5467. Epub 2012 Mar 12. PMID 22412147
- [Background] National Cancer Institute, LIVESTRONG Young Adult Alliance. Closing the Gap: Research and Care Imperatives for Adolescents and Young Adults with Cancer (Report of the Adolescent and Young Adult Oncology Progress Review Group).; 2006. https://www.livestrong.org/content/closing-gap-research-and-care-imperatives-adolescents-and-young-adults-cancer.
- [Background] Richter D, Koehler M, Friedrich M, Hilgendorf I, Mehnert A, Weissflog G. Psychosocial interventions for adolescents and young adult cancer patients: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2015 Sep;95(3):370-86. doi: 10.1016/j.critrevonc.2015.04.003. Epub 2015 Apr 16. PMID 25922217
- [Background] Chan A, Gan YX, Oh SK, Ng T, Shwe M, Chan R, Ng R, Goh B, Tan YP, Fan G. A culturally adapted survivorship programme for Asian early stage breast cancer patients in Singapore: A randomized, controlled trial. Psychooncology. 2017 Oct;26(10):1654-1659. doi: 10.1002/pon.4357. Epub 2017 Jan 25. PMID 28024163
- [Background] Lim HA, Mahendran R, Chua J, Peh CX, Lim SE, Kua EH. The Distress Thermometer as an ultra-short screening tool: a first validation study for mixed-cancer outpatients in Singapore. Compr Psychiatry. 2014 May;55(4):1055-62. doi: 10.1016/j.comppsych.2014.01.008. Epub 2014 Jan 18. PMID 24556515
- [Background] Mahendran R, Lim HA, Chua J, Lim SE, Kua EH. Psychosocial concerns of cancer patients in Singapore. Asia Pac J Clin Oncol. 2017 Apr;13(2):e96-e103. doi: 10.1111/ajco.12344. Epub 2015 Apr 9. PMID 25856735
- [Background] Watson M, Law M, Maguire B, et al. Further development of a quality of life measure for cancer patients; the Rotterdam Symptom Checklist (revised). Psychooncology. 1992;1:35-44.
- [Background] Ewing JE, King MT, Smith NF. Validation of modified forms of the PedsQL generic core scales and cancer module scales for adolescents and young adults (AYA) with cancer or a blood disorder. Qual Life Res. 2009 Mar;18(2):231-44. doi: 10.1007/s11136-008-9424-4. Epub 2009 Jan 23. PMID 19165624
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Mitchell AJ. Short screening tools for cancer-related distress: a review and diagnostic validity meta-analysis. J Natl Compr Canc Netw. 2010 Apr;8(4):487-94. doi: 10.6004/jnccn.2010.0035. PMID 20410338